CLINICAL TRIAL: NCT04136028
Title: A Retrospective Analysis of Efficacy and Safety of Interleukin-1 Receptor Inhibitor for the Treatment of Granulomatous Complications in Patients With Chronic Granulomatous Disease
Brief Title: IL-1 Receptor Inhibitor for Granulomatous Complications in Patients With Chronic Granulomatous Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2019-05
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease; Anakinra; Kineret
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention/treatment (Experimental): Anakinra (Kineret)
  Interventions: Drug: Kineret

INTERVENTIONS:
Drug: Kineret — Kineret at a dose of 8 mg/kg per day subcutaneously daily, every day at the same time
  Other Names: IL-1 receptor inhibitor

SUMMARY:
"Kineret" (INN: Anakinra) neutralizes the biological activity of interleukin-1α (IL-1α) and interleukin-1β (IL-1β) by the concurrent inhibition of binding to interleukin-1 receptor I (IL-1RI). Interleukin-1 (IL-1) is the main pro-inflammatory cytokine that mediates many cellular responses. Anakinra inhibits the reactions caused by IL-1 in vitro, including the induction of nitric oxide and prostaglandin E2 and / or the formation of collagenase by synovial cells, fibroblasts and chondrocytes. According to published data, patients with the chronic granulomatous disease have an increased secretion of interleukin-1, which contributes to the development of granulomatous inflammation. Blocking interleukin-1 reduces the activity of the main pro-inflammatory complex - the inflammasomes, and also restores the autophagy process impaired in patients with chronic granulomatous disease. In this way, inhibition of the IL-1 receptor prevents the activation of innate immunity cells and prevents the maintenance of pathological pro-inflammatory signaling in conditions of IL-1 overproduction. The efficacy and safety of therapy with the above drug is based on the results of international studies on the using of anakinra in patients with chronic granulomatous disease.

DETAILED DESCRIPTION:
The research will include a group of patients with a molecular-genetic confirmed diagnosis of chronic granulomatous disease, which has granulomatous complications on the basis of an initial comprehensive survey.

This examination will include clinical data; laboratory tests - clinical and biochemical analysis of blood (with an assessment of inflammatory activity); molecular-genetic methods for detecting mutations in the genes CYBB, CYBA, NCF2, NCF1 or NCF4; methods for studying the functional activity of neutrophils (chemiluminescence of neutrophils, test with rhodamine); methods for assessing pro-inflammatory interleukins; microbiological testing of bronchoalveolar lavage; histological studу of lung biopsies; as well as the results of visualization techniques (ultrasound investigation of the abdominal organs, CT scan of the chest and abdominal organs). Negative galactomannan and lack of microorganism growth in bronchoalveolar lavage and/or lack of response to complex antibacterial and antifungal therapy for two to three weeks confirm the presence of granulomatous complications in patients. The next step is therapy with an inhibitor of IL-1 receptor (Anakinra). Evaluation of the efficacy and safety therapy is based on the results of control examinations after 3-6 months from the start of treatment and includes an assessment of the level of C-reactive protein and pro-inflammatory cytokines, as well as the results of CT scan of the chest and abdominal organs.

ELIGIBILITY:
Inclusion Criteria:

* Granulomatous changes in the lungs or liver according to CT scan.
* Negative galactomannan and lack of microorganism growth in bronchoalveolar lavage and/or lack of response to complex antibacterial and antifungal therapy for two to three weeks.
* Signed informed consent

Exclusion Criteria:

* Patients, who do not meet the inclusion criteria.
* The reluctance of the patient or his legal representatives to participate in the research.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Estimated)
Dates: Start 2015-09-25 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 months
  Assessment of overall survival in patients with chronic granulomatous disease during therapy with an inhibitor of IL-1 receptor

SECONDARY OUTCOMES:
3 month- event-free survival | 3 months
  Assessment of event-free survival in patients with chronic granulomatous disease after treatment of granulomatous complications with an inhibitor of the IL-1 receptor (Anakinra).
6 month-event-free survival | 6 months
  Assessment of event-free survival in patients with chronic granulomatous disease after treatment of granulomatous complications with an inhibitor of the IL-1 receptor (Anakinra).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Shcherbina, PhD, Principal Investigator — National Research Center for Pediatric Hematology , Moscow, Russian Federation
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Background] van de Veerdonk FL, Dinarello CA. Deficient autophagy unravels the ROS paradox in chronic granulomatous disease. Autophagy. 2014 Jun;10(6):1141-2. doi: 10.4161/auto.28638. PMID 24879159
- [Background] de Luca A, Smeekens SP, Casagrande A, Iannitti R, Conway KL, Gresnigt MS, Begun J, Plantinga TS, Joosten LA, van der Meer JW, Chamilos G, Netea MG, Xavier RJ, Dinarello CA, Romani L, van de Veerdonk FL. IL-1 receptor blockade restores autophagy and reduces inflammation in chronic granulomatous disease in mice and in humans. Proc Natl Acad Sci U S A. 2014 Mar 4;111(9):3526-31. doi: 10.1073/pnas.1322831111. Epub 2014 Feb 18. PMID 24550444
- [Background] Hahn KJ, Ho N, Yockey L, Kreuzberg S, Daub J, Rump A, Marciano BE, Quezado M, Malech HL, Holland SM, Heller T, Zerbe CS. Treatment With Anakinra, a Recombinant IL-1 Receptor Antagonist, Unlikely to Induce Lasting Remission in Patients With CGD Colitis. Am J Gastroenterol. 2015 Jun;110(6):938-9. doi: 10.1038/ajg.2015.135. No abstract available. PMID 26052777
- [Background] Meissner F, Seger RA, Moshous D, Fischer A, Reichenbach J, Zychlinsky A. Inflammasome activation in NADPH oxidase defective mononuclear phagocytes from patients with chronic granulomatous disease. Blood. 2010 Sep 2;116(9):1570-3. doi: 10.1182/blood-2010-01-264218. Epub 2010 May 21. PMID 20495074